CLINICAL TRIAL: NCT05447819
Title: Migration and Functional Outcome of DELTA Xtend Reverse Shoulder Lateralized Glenosphere Line Extension System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Principal Investigator, Marie Louise Jensen, Principal investigator, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-21042181
Record Dates: First submitted 2022-06-24; First posted 2022-07-07 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Rotator Cuff Arthropathy or Degeneration of the Glenohumeral Joint with Severe Posterior Wear

STUDY DESIGN:
Intervention Model Description: Based on the sample calculation the investigators intend to include a total number of 122 patients of which the first 56 patients will be studied using MB-RSA and DXA. The patients are allocated into two groups of equal of size:
  1. DELTA Xtend Reverse Shoulder System Lateralized Glenosphere Line Extension (intervention group)
  2. Standard DELTA Xtend Reverse Shoulder System (control group).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: It is not possible to blind the observer when implant migration is evaluated using RSA. The patient-reported outcomes are solely evaluated by the patients before the follow-up examination without involving surgeons or observer
  Blinding of the patients:
  The patients will be blinded to their allocated treatment the first two years after surgery.
  Blinding of Statistician:
  The randomization is blinded to the statistician who perform the analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DELTA Xtend Reverse Shoulder System Lateralized Glenosphere Line Extension (Experimental): By using a lateralized glensphere complications can be reduced and patients can achieve an improved outcome.
  Currently, little is known about the results of the lateralized design. The initial results have been promising, but migration and eventually loosening of the prosthesis can lead to poor results and, in some cases, revision
  Interventions: Procedure: Reverse shoulder arthroplsaty
- Standard DELTA Xtend Reverse Shoulder System (Active Comparator): A design with a standard glenosphere is currently regarded as the standard treatment
  Interventions: Procedure: Reverse shoulder arthroplsaty

INTERVENTIONS:
Procedure: Reverse shoulder arthroplsaty — Patients with the diagnosis of rotator cuff arthropathy (degeneration of the glenohumeral joint and wear or tear of at least one rotator cuff tendon) or degeneration of the glenohumeral joint with severe posterior wear with an indication of a reverse total shoulder arthroplasty

SUMMARY:
This is a randomized controlled trial comparing the DELTA Xtend Reverse Shoulder System Lateralized Glenosphere Line Extension (intervention group) with the standard DELTA Xtend Reverse Shoulder System (control group). All Danish citizens with rotator cuff arthropathy or degeneration of the glenohumeral joint with severe posterior wear indicating a reverse total shoulder arthroplasty referred to the orthopedic department at Herlev and Gentofte Hospital, Copenhagen University Hospital will be considered for participation in the trial. The following exclude from participation in the study: Below 50 years of age; Cognitive or linguistic impairment; insufficient glenoid bone stock; previous fracture in the upper extremities; autoimmune mediated inflammatory arthritis.A total of 122 patients will be included of which 56 will be part of the roentgen radiostereometric analysis. This will allow a maximum of 20% drop out. The primary outcome is magnitude and pattern of migration of the glenoid component and functional outcome by Western Ontario Osteoarthritis of the Shoulder Index (WOOS score). The secondary outcomes are position of arthroplasty, loosening, inferior scapular notching, patient-reported outcomes, functional outcome, readmission, complications, revisions, changes in bone mineral density of the proximal humerus assessed by duel energy x-ray absorptiometry and economy (cost utility analysis). The patients are examined before the operation and 1 week and 3, 6, 12 and 24 months after the operation.

ELIGIBILITY:
Inclusion Criteria:

1. Rotator cuff arthropathy defined as degeneration of the glenohumeral joint and wear or tear of at least one rotator cuff tendon
2. Degeneration of the glenohumeral joint with intact rotator cuff function but severe posterior wear of the glenoid (>20 degrees posterior wear)
3. Insufficient effect of non-surgical treatment with symptoms severe enough to justify shoulder arthroplasty.
4. ASA (American Society of Anesthesiology) score 1-3, physically fit for surgery and rehabilitation

Exclusion Criteria:

1. Below 50 years of age
2. Cognitive or linguistic impairment
3. Insufficient glenoid bone-stock
4. Previous fracture in the upper extremities
5. Patients with autoimmune mediated inflammatory arthritis
6. Glenoid border medial to the medial border of the coracoid on a true AP radiograph

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Radiostereometric analysis (RSA) [ Time Frame: Change from 1 week postoperatively to 3 months, 6 months, and at 1 and 2 years postoperatively ] | At 1 week and at 3 months, 6 months, 1 year and 2 years
  A special x-ray examination technique based upon insertion of small metal beads into the bone surrounding an implant and attachment of beads to the prosthesis (or using 3-dimensional models of the implant (CAD models) = model-based RSA (MB-RSA)). In this way, implant migration can be measured extremely accurate.
Western Ontario Osteoarthritis of the Shoulder index (WOOS) [ Time Frame: Change in WOOS score from preoperatively to 3 months, 6 months, and at 1 and 2 years postoperatively ] | preoperatively and at at 3 months, 6 months, 1 year and 2 years
  The WOOS is a disease-specific patient-reported outcome (Lo IK et al 2001). There are 19 questions divided into four domains: Physical symptoms, sports and work, lifestyle and emotions. Each question is answered on a visual analogue scale ranging from 0 to 100. The overall score ranges from 0 to 1900, with 1900 being the worst. For ease of interpretation, the scores are converted to a percentage of the maximum score. There will be used a Danish version of WOOS (Rasmussen JV et al 2013) which was translated according to the guidelines of Guillemin, Bombardier and Beaton (Guillemin F et al 1993). It was validated with classical test theory in a cohort of patients treated with shoulder arthroplasty for osteoarthritis.

SECONDARY OUTCOMES:
Plain radiographs [ Time Frame: Preoperatively and at 1 week, 3 months and at 1 and 2 years postoperatively ] | Preoperatively and at 1 week, 3 months and at 1 and 2 years postoperatively
  There will be used an anterior-posterior and a lateral view. The radiographs are used to evaluate the position of the component and to evaluate loosening as the cause of failure.
Duel energy x-ray absorptiometry (DXA) [ Time Frame: Preoperatively and at 1 week, 3 months, 6 months, and at 1 and 2 years postoperatively ] | Preoperatively and at 1 week, 3 months, 6 months, and at 1 and 2 years postoperatively
  Changes in bone mineral density (BMD) in close relation to an orthopedic implant can be measured by duel x-ray absorptiometry (DXA)
Constant-Murley score [ Time Frame: Preoperatively and 3 months, 6 months, and at 1 and 2 years postoperatively ] | Preoperatively and 3 months, 6 months, and at 1 and 2 years postoperatively
  The Constant-Murley Score includes an assessment of: pain; activities of daily living (ADL); range of motion; and strength. There are a possible 35 points given for the subjective assessment of pain and the ability to perform ADL. There are a possible 65 points given for an objective assessment, of which 40 points are allocated to range of motion and 25 points are allocated to strength. The maximum of 100 point indicates a shoulder with no disability. There will be used a Danish version (Ban I et al 2013) of the modified score described by Con¬stant and colleagues in 2008 (Constant CR et al 2008).
Oxford Shoulder Score (OSS) [ Time Frame: Preoperatively and 3 months, 6 months, and at 1 and 2 years postoperatively ] | Preoperatively and 3 months, 6 months, and at 1 and 2 years postoperatively
  Oxford Shoulder Score (OSS): The OSS was conceived as a measurement tool for the assessment of pain and function after elective shoulder surgery (Dawson J et al 1996). There are 12 questions with each item scored from 1-5. The overall score ranges from 12 to 60, with 60 being the worst. For ease of interpretation, the scores are converted to a percentage of the maximum score. There will be used a Danish version of OSS which was translated and validated with classical test theory (Frich LH et al 2011).
Side effects and complications [ Time Frame: 2 years postoperatively ] | 2 years postoperatively
  There will be recorded any case of medical complications (embolism, cardiovascular event, pneumonia) and complications related to the surgical procedure (fractures, nerve injuries, deep and superficial infections, malpositioning of the components, instability, and dislocation) and revisions defined by removal or exchange of any component.
Pain and patient-satisfaction: visual analogue scale (VAS) [ Time Frame: 3 months, 6 months, and at 1 and 2 years postoperatively ] | 3 months, 6 months, and at 1 and 2 years postoperatively
  Pain is answered on a visual analogue scale (VAS) ranging from 0 to 10, with 10 being the worst. Patients are asked to categorize the result as excellent, very good, good, fair and poor.
Cost-utility analysis [ Time Frame: 2 years postoperatively ] | 2 years postoperatively
  In modern health economics, thresholds have been estimated for acceptable cost-utility ratios - the threshold for how much health care providers will pay for an extra quality- adjusted life year (QALY). In England and in Europe, the threshold for an extra QALY is set at 20,000-30,000 pounds and 30,000 Euros respectively. The cost utility of the Comprehensive Nano stemless shoulder arthroplasty will be compared with these thresholds and with the cost utility of the uncemented Comprehensive stemmed total shoulder arthroplasty. The EQ-5D will be used to estimate QALY for individual patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev and Gentofte Hospital, Hellerup, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andersen MR, Winther NS, Lind T, Schroder HM, Flivik G, Petersen MM. Low Preoperative BMD Is Related to High Migration of Tibia Components in Uncemented TKA-92 Patients in a Combined DEXA and RSA Study With 2-Year Follow-Up. J Arthroplasty. 2017 Jul;32(7):2141-2146. doi: 10.1016/j.arth.2017.02.032. Epub 2017 Feb 28. PMID 28410836
- [Background] Andersen MR, Winther N, Lind T, SchroDer H, Flivik G, Petersen MM. Monoblock versus modular polyethylene insert in uncemented total knee arthroplasty. Acta Orthop. 2016 Dec;87(6):607-614. doi: 10.1080/17453674.2016.1233654. Epub 2016 Sep 20. PMID 27649258
- [Background] Andersen MR, Winther NS, Lind T, Schroder HM, Mork Petersen M. Bone Remodeling of the Distal Femur After Uncemented Total Knee Arthroplasty-A 2-Year Prospective DXA Study. J Clin Densitom. 2018 Apr-Jun;21(2):236-243. doi: 10.1016/j.jocd.2017.05.001. Epub 2017 Sep 13. PMID 28918227
- [Background] ten Broeke RH, Hendrickx RP, Leffers P, Jutten LM, Geesink RG. Randomised trial comparing bone remodelling around two uncemented stems using modified Gruen zones. Hip Int. 2012 Jan-Feb;22(1):41-9. doi: 10.5301/HIP.2012.9103. PMID 22383318
- [Background] Constant CR, Gerber C, Emery RJ, Sojbjerg JO, Gohlke F, Boileau P. A review of the Constant score: modifications and guidelines for its use. J Shoulder Elbow Surg. 2008 Mar-Apr;17(2):355-61. doi: 10.1016/j.jse.2007.06.022. Epub 2008 Jan 22. No abstract available. PMID 18218327
- [Background] Dawson J, Fitzpatrick R, Carr A. Questionnaire on the perceptions of patients about shoulder surgery. J Bone Joint Surg Br. 1996 Jul;78(4):593-600. PMID 8682827
- [Background] Denard PJ, Walch G. Current concepts in the surgical management of primary glenohumeral arthritis with a biconcave glenoid. J Shoulder Elbow Surg. 2013 Nov;22(11):1589-98. doi: 10.1016/j.jse.2013.06.017. Epub 2013 Sep 3. PMID 24007651
- [Background] Frich LH, Noergaard PM, Brorson S. Validation of the Danish version of Oxford Shoulder Score. Dan Med Bull. 2011 Nov;58(11):A4335. PMID 22047932
- [Background] Friedman RJ, Barcel DA, Eichinger JK. Scapular Notching in Reverse Total Shoulder Arthroplasty. J Am Acad Orthop Surg. 2019 Mar 15;27(6):200-209. doi: 10.5435/JAAOS-D-17-00026. PMID 30260909
- [Background] Gluer CC, Steiger P, Selvidge R, Elliesen-Kliefoth K, Hayashi C, Genant HK. Comparative assessment of dual-photon absorptiometry and dual-energy radiography. Radiology. 1990 Jan;174(1):223-8. doi: 10.1148/radiology.174.1.2294552.
- [Background] Guillemin F, Bombardier C, Beaton D. Cross-cultural adaptation of health-related quality of life measures: literature review and proposed guidelines. J Clin Epidemiol. 1993 Dec;46(12):1417-32. doi: 10.1016/0895-4356(93)90142-n. PMID 8263569
- [Background] Henninger HB, Barg A, Anderson AE, Bachus KN, Burks RT, Tashjian RZ. Effect of lateral offset center of rotation in reverse total shoulder arthroplasty: a biomechanical study. J Shoulder Elbow Surg. 2012 Sep;21(9):1128-35. doi: 10.1016/j.jse.2011.07.034. Epub 2011 Oct 29. PMID 22036546
- [Background] Jensen CL, Petersen MM, Schroder HM, Flivik G, Lund B. Revision total knee arthroplasty with the use of trabecular metal cones: a randomized radiostereometric analysis with 2 years of follow-up. J Arthroplasty. 2012 Dec;27(10):1820-1826.e2. doi: 10.1016/j.arth.2012.04.036. Epub 2012 Jul 13. PMID 22795879
- [Background] Jensen CL, Petersen MM, Schroder HM, Lund B. Bone mineral density changes of the proximal tibia after revision total knee arthroplasty. A randomised study with the use of porous tantalum metaphyseal cones. Int Orthop. 2012 Sep;36(9):1857-63. doi: 10.1007/s00264-012-1601-y. Epub 2012 Jun 26. PMID 22733440
- [Background] Karrholm J, Gill RH, Valstar ER. The history and future of radiostereometric analysis. Clin Orthop Relat Res. 2006 Jul;448:10-21. doi: 10.1097/01.blo.0000224001.95141.fe. PMID 16826090
- [Background] Karrholm J. Radiostereometric analysis of early implant migration - a valuable tool to ensure proper introduction of new implants. Acta Orthop. 2012 Dec;83(6):551-2. doi: 10.3109/17453674.2012.745352. Epub 2012 Nov 5. No abstract available. PMID 23126576
- [Background] Laursen MB, Nielsen PT, Soballe K. Bone remodelling around HA-coated acetabular cups : a DEXA study with a 3-year follow-up in a randomised trial. Int Orthop. 2007 Apr;31(2):199-204. doi: 10.1007/s00264-006-0148-1. Epub 2006 Jun 8. PMID 16761153
- [Background] Lawrence C, Williams GR, Namdari S. Influence of Glenosphere Design on Outcomes and Complications of Reverse Arthroplasty: A Systematic Review. Clin Orthop Surg. 2016 Sep;8(3):288-97. doi: 10.4055/cios.2016.8.3.288. Epub 2016 Aug 10. PMID 27583112
- [Background] Lo IK, Griffin S, Kirkley A. The development of a disease-specific quality of life measurement tool for osteoarthritis of the shoulder: The Western Ontario Osteoarthritis of the Shoulder (WOOS) index. Osteoarthritis Cartilage. 2001 Nov;9(8):771-8. doi: 10.1053/joca.2001.0474. PMID 11795997
- [Background] Marchetti ME, Houde JP, Steinberg GG, Crane GK, Goss TP, Baran DT. Humeral bone density losses after shoulder surgery and immobilization. J Shoulder Elbow Surg. 1996 Nov-Dec;5(6):471-6. doi: 10.1016/s1058-2746(96)80020-6. PMID 8981273
- [Background] Mazess RB, Barden HS. Measurement of bone by dual-photon absorptiometry (DPA) and dual-energy X-ray absorptiometry (DEXA). Ann Chir Gynaecol. 1988;77(5-6):197-203. PMID 3076046
- [Background] Mechlenburg I, Klebe TM, Dossing KV, Amstrup A, Soballe K, Stilling M. Evaluation of periprosthetic bone mineral density and postoperative migration of humeral head resurfacing implants: two-year results of a randomized controlled clinical trial. J Shoulder Elbow Surg. 2014 Oct;23(10):1427-36. doi: 10.1016/j.jse.2014.05.012. PMID 25220196
- [Background] Mollon B, Mahure SA, Roche CP, Zuckerman JD. Impact of scapular notching on clinical outcomes after reverse total shoulder arthroplasty: an analysis of 476 shoulders. J Shoulder Elbow Surg. 2017 Jul;26(7):1253-1261. doi: 10.1016/j.jse.2016.11.043. Epub 2017 Jan 19. PMID 28111179
- [Background] Nelissen RG, Pijls BG, Karrholm J, Malchau H, Nieuwenhuijse MJ, Valstar ER. RSA and registries: the quest for phased introduction of new implants. J Bone Joint Surg Am. 2011 Dec 21;93 Suppl 3:62-5. doi: 10.2106/JBJS.K.00907. PMID 22262426
- [Background] Nuttall D, Haines JF, Trail IA. The early migration of a partially cemented fluted pegged glenoid component using radiostereometric analysis. J Shoulder Elbow Surg. 2012 Sep;21(9):1191-6. doi: 10.1016/j.jse.2011.07.028. Epub 2011 Nov 1. PMID 22047783
- [Background] Nuttall D, Birch A, Haines JF, Trail IA. Radiostereographic analysis of a shoulder surface replacement: does hydroxyapatite have a place? Bone Joint J. 2014 Aug;96-B(8):1077-81. doi: 10.1302/0301-620X.96B8.30534. PMID 25086124
- [Background] Nuttall D, Haines JF, Trail II. A study of the micromovement of pegged and keeled glenoid components compared using radiostereometric analysis. J Shoulder Elbow Surg. 2007 May-Jun;16(3 Suppl):S65-70. doi: 10.1016/j.jse.2006.01.015. Epub 2006 Aug 7. PMID 17493557
- [Background] Rasmussen JV, Jakobsen J, Olsen BS, Brorson S. Translation and validation of the Western Ontario Osteoarthritis of the Shoulder (WOOS) index - the Danish version. Patient Relat Outcome Meas. 2013 Sep 18;4:49-54. doi: 10.2147/PROM.S50976. eCollection 2013. PMID 24133377
- [Background] Rasmussen JV, Olsen BS, Sorensen AK, Hrobjartsson A, Brorson S. Resurfacing hemiarthroplasty compared to stemmed hemiarthroplasty for glenohumeral osteoarthritis: a randomised clinical trial. Int Orthop. 2015 Feb;39(2):263-9. doi: 10.1007/s00264-014-2505-9. Epub 2014 Aug 27. PMID 25159010
- [Background] Rasmussen JV, Hole R, Metlie T, Brorson S, Aarimaa V, Demir Y, Salomonsson B, Jensen SL. Anatomical total shoulder arthroplasty used for glenohumeral osteoarthritis has higher survival rates than hemiarthroplasty: a Nordic registry-based study. Osteoarthritis Cartilage. 2018 May;26(5):659-665. doi: 10.1016/j.joca.2018.02.896. Epub 2018 Feb 21. PMID 29474992
- [Background] Rasmussen JV, Olsen BS, Al-Hamdani A, Brorson S. Outcome of Revision Shoulder Arthroplasty After Resurfacing Hemiarthroplasty in Patients with Glenohumeral Osteoarthritis. J Bone Joint Surg Am. 2016 Oct 5;98(19):1631-1637. doi: 10.2106/JBJS.15.00934. PMID 27707849
- [Background] Rasmussen JV, Polk A, Brorson S, Sorensen AK, Olsen BS. Patient-reported outcome and risk of revision after shoulder replacement for osteoarthritis. 1,209 cases from the Danish Shoulder Arthroplasty Registry, 2006-2010. Acta Orthop. 2014 Apr;85(2):117-22. doi: 10.3109/17453674.2014.893497. PMID 24650020
- [Background] Rasmussen JV, Polk A, Sorensen AK, Olsen BS, Brorson S. Outcome, revision rate and indication for revision following resurfacing hemiarthroplasty for osteoarthritis of the shoulder: 837 operations reported to the Danish Shoulder Arthroplasty Registry. Bone Joint J. 2014 Apr;96-B(4):519-25. doi: 10.1302/0301-620X.96B4.31850. PMID 24692621
- [Background] Roche CP, Stroud NJ, Martin BL, Steiler CA, Flurin PH, Wright TW, DiPaola MJ, Zuckerman JD. The impact of scapular notching on reverse shoulder glenoid fixation. J Shoulder Elbow Surg. 2013 Jul;22(7):963-70. doi: 10.1016/j.jse.2012.10.035. Epub 2013 Jan 16. PMID 23333170
- [Background] Ryd L, Albrektsson BE, Carlsson L, Dansgard F, Herberts P, Lindstrand A, Regner L, Toksvig-Larsen S. Roentgen stereophotogrammetric analysis as a predictor of mechanical loosening of knee prostheses. J Bone Joint Surg Br. 1995 May;77(3):377-83. PMID 7744919
- [Background] Sirveaux F, Favard L, Oudet D, Huquet D, Walch G, Mole D. Grammont inverted total shoulder arthroplasty in the treatment of glenohumeral osteoarthritis with massive rupture of the cuff. Results of a multicentre study of 80 shoulders. J Bone Joint Surg Br. 2004 Apr;86(3):388-95. doi: 10.1302/0301-620x.86b3.14024. PMID 15125127
- [Background] Stilling M, Mechlenburg I, Amstrup A, Soballe K, Klebe T. Precision of novel radiological methods in relation to resurfacing humeral head implants: assessment by radiostereometric analysis, DXA, and geometrical analysis. Arch Orthop Trauma Surg. 2012 Nov;132(11):1521-30. doi: 10.1007/s00402-012-1580-x. Epub 2012 Jul 7. PMID 22773108
- [Background] Ten Brinke B, Beumer A, Koenraadt KLM, Eygendaal D, Kraan GA, Mathijssen NMC. The accuracy and precision of radiostereometric analysis in upper limb arthroplasty. Acta Orthop. 2017 Jun;88(3):320-325. doi: 10.1080/17453674.2017.1291872. Epub 2017 Mar 2. PMID 28464752
- [Background] Trozzi C, Kaptein BL, Garling EH, Shelyakova T, Russo A, Bragonzoni L, Martelli S. Precision assessment of model-based RSA for a total knee prosthesis in a biplanar set-up. Knee. 2008 Oct;15(5):396-402. doi: 10.1016/j.knee.2008.05.001. Epub 2008 Jul 16. PMID 18635360
- [Background] Valstar ER, Gill R, Ryd L, Flivik G, Borlin N, Karrholm J. Guidelines for standardization of radiostereometry (RSA) of implants. Acta Orthop. 2005 Aug;76(4):563-72. doi: 10.1080/17453670510041574. PMID 16195075
- [Background] Valstar E, Kaptein B, Nelissen R. Radiostereometry and new prostheses. Acta Orthop. 2012 Apr;83(2):103-4. doi: 10.3109/17453674.2012.678796. Epub 2012 Apr 11. No abstract available. PMID 22489889
- [Background] Winther NS, Jensen CL, Jensen CM, Lind T, Schroder HM, Flivik G, Petersen MM. Comparison of a novel porous titanium construct (Regenerex(R)) to a well proven porous coated tibial surface in cementless total knee arthroplasty - A prospective randomized RSA study with two-year follow-up. Knee. 2016 Dec;23(6):1002-1011. doi: 10.1016/j.knee.2016.09.010. Epub 2016 Oct 19. PMID 27769563
- [Background] Winther N, Jensen C, Petersen M, Lind T, Schroder H, Petersen M. Changes in bone mineral density of the proximal tibia after uncemented total knee arthroplasty. A prospective randomized study. Int Orthop. 2016 Feb;40(2):285-94. doi: 10.1007/s00264-015-2852-1. Epub 2015 Jul 17. PMID 26183139